CLINICAL TRIAL: NCT05545007
Title: Phase III Randomized Trial Comparing Preoperative Hypofractionated Radiosurgery (HSRS) to Postoperative Hypofractionated Radiosurgery (HSRS) for Patients With Large Brain Metastases (= 2.1cm) Suitable for Surgical Resection
Brief Title: Preoperative vs Postoperative Hypofractionated Radiosurgery for Patients With Large Brain Metastases
Acronym: SUPPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Brainlab AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3270
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases, Adult
Keywords: pre-operative hypofractionated radiosurgery; surgical resection; large brain metastases; post-operative hypofractionated radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSRS pre-operative (Experimental): Patients undergo HSRS (hypofractionated Radiosurgery) on day 1, consisting in 27 Gray (gy) administered in 3 daily fractions.
  Within 1 weeks, patients undergo surgical resection.
  Interventions: Radiation: Hypofractionated Radiosurgery (HSRS); Procedure: Brain metastases surgical resection
- HSRS post-operative (Active Comparator): Patients undergo surgical resection on day 1. Within 4-6 weeks, patients undergo HSRS (hypofractionated Radiosurgery), consisting in 27 Gray (gy) administered in 3 daily fractions.
  Interventions: Radiation: Hypofractionated Radiosurgery (HSRS); Procedure: Brain metastases surgical resection

INTERVENTIONS:
Radiation: Hypofractionated Radiosurgery (HSRS) — HSRS converges multiple radiation beams to deliver a single, large dose of radiation to a discrete tumor target with high precision, thereby minimizing radiation dose to the surrounding normal tissue.
Procedure: Brain metastases surgical resection — Complete surgical resection of brain lesions with adeguate margins.

SUMMARY:
This is a phase III randomized trial with the aim to compare preoperative HSRS to postoperative HSRS in patients with large at least one BMs from solid tumors suitable for surgical resection.

DETAILED DESCRIPTION:
The occurrence of BMs is a huge and challenging issue affecting about 20-40% of patients with solid primary tumors. Among these, about 25% of patients harbored large BMs, defined as ≥ 2.1 cm. Single dose SRS, using the dose guidelines suggested by the Radiation Therapy Oncology Group (RTOG) 90-05 study, obtains an unsatisfactory local control (LC) rate ranging from 45-49%. In this subset of patients other treatment pathways have been investigated. In the 1990s, Patchell and colleagues determined that patients with good functional status, and solitary intracranial metastases should undergo surgical resection. Unfortunately, surgery alone is able to control tumor in only 50% of patients, and an adjuvant radiation therapy (RT) is required. For several years, adjuvant whole brain radiation therapy (WBRT) has been considered the standard of cure, but a high risk of impairment in neurological functions was recorded, without an actual benefit on survival. Different RT approaches have been inquired with the aim to reduce neurological toxicity preserving the same brain tumor control. Recent randomized trials showed that single dose SRS on the tumor bed might be a valid, and less toxic alternative to WBRT, although an increased risk of radio necrosis (RN) was noticed when large surgical cavities are treated. In the last years hypofractionated stereotactic radiosurgery (HSRS) has gained interest. Its goal is to reduce the risk of RN compared to single dose SRS, while providing similar, or perhaps, improved LC, probably in relation to the need of reducing the dose prescribed in cases of larger lesions using SRS.

However, there has been increasing evidence that patients treated with postoperative SRS have an increased rates of leptomeningeal disease (LMD) occurrence than what was observed when postoperative WBRT was used as the standard. Several retrospective studies have demonstrated a LMD rates up to 31% in the postoperative SRS setting.

The proposed mechanism of this increased risk is iatrogenic tumor dissemination into the cerebrospinal fluid (CSF) at the time of surgical resection, which was not as apparent when the entire intracranial CSF space was treated with routine postoperative WBRT, but has become more apparent with increasing use of postoperative SRS only. It is important to note that a standardized definition of radiographic LMD does not exist and ascertainment bias as to what constitutes radiographic LMD (vs local or distant meningeal failure as an example) is an unresolved issue.

Due to the perceived drawbacks of postoperative SRS, namely the need for cavity margin expansion due to target delineation uncertainty, the variable postoperative clinical course and potential delay in administering postoperative SRS, and the theoretical risk of tumor spillage into CSF at the time of surgery, investigators began to study the use of preoperative SRS as an alternative paradigm to maximize local control of the resection cavity and minimize neurocognitive detriment associated with WBRT. Preoperative SRS has several potential advantages compared to postoperative SRS consisting in :

* a better target delineation to an intact lesion
* the reduction of normal brain irradiated considering the useless of additional margins
* the potential prevention of any cells spilled during resection
* a greater oxygenation ratio of the intact region
* a sterilization effect
* the resection of the majority of irradiated tissues Based on this background we designed this phase III randomized trial comparing preoperative HSRS to postoperative HSRS in patients with large at least one BMs from solid tumors suitable for surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histological or cytological or radiological confirmation of solid tumor malignancy
* Clinical indication for surgical resection of one brain metastasis
* Karnosky performance status (KPS) ≥70
* Controlled or responsive extra cranial metastatic lesions
* Limited brain metastases (1-4 BMs)
* Single metastatic lesion ≥ 2.1 cm in maximum diameter (4 cm3)
* Lesions ≤2 cm conditioning mass effect or neurological deficits or massive edema unresponsive to steroids
* Written informed consent form

Exclusion Criteria:

* Prior WBRT
* KPS < 70
* Diagnosis of small cell lung cancer (SCLC), germinal cell tumour or Lymphoproliferative disease
* Pregnant women
* Prior open neurosurgery for malignancy
* More than 4 brain metastases
* Patients with incompatibility to perform MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of LMD (leptomeningeal disease) occurrence | 1 year
  Rate of LMD occurrence in patients who receive HSRS prior to surgery as compared to patients who receive HSRS after surgery. This assessment will be evaluated through radiological images.

SECONDARY OUTCOMES:
Rate of local recurrence | 1 year
  To evaluate for patients undergone pre-operative as compared to post-operative HSRS whether there is a decreased rate of local recurrence. This assessment will be evaluated through radiological images.
Rate of brain distant progression | 1 year
  To evaluate for patients undergone pre-operative as compared to post-operative HSRS whether there is a decreased rate of brain distant progression. This assessment will be evaluated through radiological images.
Overall Survival | 1 year
  To evaluate for patients with brain metastases whether there is improved overall survival for patients who receive HSRS prior to surgery as compared to patients who receive HSRS after surgery.
Radiation Necrosis Evaluation | 1 year
  To evaluate for patients undergone pre-operative as compared to post-operative HSRS whether there is a decreased rate of symptomatic radiation necrosis (RN). RN will be evaluated through radiological images.
Rate of surgical Morbidity | 1 year
  To evaluate whether preoperative SRS increases rates of surgical morbidity including postoperative complications such as wound infection, need for longer hospital stays, readmission and eventual delay of systemic treatments
Quality of Life and neurocognitive functions evaluation | 1 year
  To evaluate quality of life (EORTC QLQ-C30, version 3.0) and neurocognitive functions throught specific questionnaires administered to patients.
  Neurocognitive test:
  * Token Test (Spinnler e Tognoni, 1987)
  * Picture naming of objects (Catricalà 2012) and of actions (Papagno et al., 2020)
  * Verbal fluency on phonemic and semantic cue (Novelli et al., 1986)
  * Rey's 15 words auditory learning test (Carlesimo et al.,1996)
  * Reproduction of the Rey figure (Caffarra et al., 2002)
  * Stroop test (Caffarra et al. 2002)
  * Trail making test (Giovagnoli et al. 1996)
  * Copy of Rey Figure (Cafarra et al., 2002)

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - ASST Spedali Civili di Brescia, Brescia, Brescia
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Florence
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milan
  - Ospedale del Mare, Naples, naples
  - Policlinico Umberto I, Rome, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Rome
  - AOU Sant'Andrea, Rome, Rome
  - Azienda Ospedaliera Santa Maria di Terni, Terni, Terni

IPD SHARING:
Plan to Share IPD: Yes